CLINICAL TRIAL: NCT06321341
Title: Open-label, Multicenter, Randomized Controlled Phase 4 Trial Evaluating the Efficacy and Safety of Vespireit, Prolonged-release Tablets (Valenta Pharm JSC, Russia) Versus Arlevert, Tablets (Menarini International Operations Luxembourg S.A., Luxembourg) in Patients With Autonomic Dysfunction Syndrome Accompanied by Functional Vertigo.
Brief Title: Efficacy and Safety of Vespireit, Prolonged-release Tablets, in Patients With Autonomic Dysfunction Syndrome Accompanied by Functional Vertigo
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Valenta Pharm JSC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BUSP-04-04-2023
Record Dates: First submitted 2024-03-13; First posted 2024-03-20 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Vertigo; Autonomic Dysfunction
MeSH Terms: conditions — Vertigo; Primary Dysautonomias | interventions — cinnarizine, dimenhydrinate drug combination

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vespireit, prolonged-release tablets, 15 mg (Experimental): Dosage regimen: 1 tablet once a day at approximately the same time in the morning under fed conditions for 28 days. The drug is taken orally, whole, without breaking and not chewing.
  Interventions: Drug: Vespireit
- Arlevert, tablets, 40 mg + 20 mg (Active Comparator): Dosage regimen: 1 tablet 3 times a day at approximately the same time under fed conditions for 28 days. The drug is taken orally, whole, without breaking and not chewing.
  Interventions: Drug: Arlevert

INTERVENTIONS:
Drug: Vespireit — Buspirone
  Arms: Vespireit, prolonged-release tablets, 15 mg
Drug: Arlevert — Dimenhydrinate + Cinnarizine
  Arms: Arlevert, tablets, 40 mg + 20 mg

SUMMARY:
This study aims to evaluate the efficacy and safety of Vespireit, prolonged-release tablets, 15 mg (Valenta Pharm JSC, Russia) in comparison with Arlevert, tablets, 40 mg + 20 mg (Menarini International Operations Luxembourg S.A., Luxembourg) in patients with autonomic dysfunction syndrome accompanied by functional vertigo.

ELIGIBILITY:
Inclusion Criteria:

1. Patient signed and dated the Informed Consent Form.
2. Males and females ≥18 to ≤ 65 years of age inclusive at the time of signing the Informed Consent Form.
3. Clinical diagnosis: G90.8 Other disorders of autonomic nervous system or G90.9 Disorder of autonomic nervous system, unspecified.
4. Diagnosed chronic functional vertigo per Barani Society criteria: total DHI score ≥ 31 points; mean MVS score ≥ 1.5 points.
5. For women of childbearing potential, a negative pregnancy test and consent to use an authorized method of contraception throughout the entire period of study participation, starting from Visit 0, and for 3 weeks after the end of the study; for men, consent to use an authorized method of contraception throughout the entire period of study participation and for 3 weeks after the end of the study.

The authorized contraceptive methods in this study are: intrauterine device, barrier method, or dual barrier method (condom or occlusive cap (diaphragm or cervical/vaginal cap) plus spermicide)). Hormonal contraception was not permitted due to insufficient data on drug interactions of buspirone.

Postmenopausal women (≥2 years of amenorrhea) or women who are surgically sterile (hysterectomy, bilateral ovariectomy, tubal ligation)) and men with documented infertility or vasectomy will also be eligible for the study.

Non-inclusion Criteria:

1. Known or suspected hypersensitivity to the active substance or any of the excipients of the investigational drugs.
2. Lactose intolerance, lactase deficiency, glucose-galactose malabsorption.
3. A cumulative score > 2 on the Suicide Risk Assessment Scale (SRAS).
4. Chronic heart failure III-IV functional classes according to the New York Heart Association (NYHA) classification, angina pectoris III-IV functional classes.
5. Presence of uncompensated peripheral vestibular hyporeflexia due to previous vestibular neuronitis, labyrinthitis, labyrinth trauma.
6. Presence at the time of screening of exacerbation of vestibular diseases with episodic vestibular syndrome.
7. Meniere's disease.
8. Established diagnosis of bilateral vestibular insufficiency.
9. Syncopal and presyncopal conditions at the time of screening.
10. Acute cardiovascular disease or surgical interventions (myocardial infarction, angioplasty, aortocoronary/mammary coronary heart bypass, unstable angina, and others) less than 6 months prior to the date of the Screening Visit.
11. Acute cerebral circulatory disorders and/or transient ischemic attacks less than 6 months prior to the date of the Screening Visit.
12. Hemodynamically significant cardiac rhythm and conduction abnormalities, including a history of cardiac rhythm and conduction abnormalities.
13. An installed artificial pacemaker.
14. Clinically significant ECG abnormalities;
15. Established diagnosis of liver failure, including history and/or altered laboratory values: increase in aspartateaminotransferase (AST), alanineaminotransferase (ALT) more than 2.5 times relative to the upper limit of normal, increase in total bilirubin more than 1.5 times above the upper limit of normal;
16. Established diagnosis of renal failure of any severity and/or creatinine clearance calculated by the Cockcroft-Gault formula at screening < 80 ml/min in women and < 90 ml/min in men.
17. Pyloroduodenal obstruction based on history.
18. Prostatic hyperplasia.
19. Thyroid function disorder according to examination and clinical and laboratory tests.
20. Parkinson's disease according to anamnesis.
21. Severe ischemic heart disease.
22. Uncontrolled hypertension with systolic blood pressure > 180 mm Hg and/or diastolic blood pressure > 110 mm Hg, or blood pressure (BP) at screening ≥140/90 or ≤ 100/60 mm Hg.
23. Uncontrolled diabetes mellitus, diabetes mellitus in decompensation.
24. Myasthenia gravis.
25. Closed-angle glaucoma.
26. Suspicion of elevated intraocular pressure at the time of screening.
27. Systemic connective tissue diseases.
28. Autoimmune diseases.
29. History or suspected elevated intracranial pressure.
30. Urinary retention due to a history of urethral and/or prostate disease.
31. Need for surgical and/or endovascular treatment in the next 15 months.
32. Epilepsy or convulsive seizures, including history of seizures.
33. Alcoholism, drug dependence, substance abuse in the history and/or at the time of screening (alcoholism - use of more than 30 ml of ethyl alcohol per day during the last 6 months; drug dependence - use of any narcotic substances in any doses during the last 6 months; substance abuse - use of any psychoactive substances in any doses during the last 6 months).
34. History of schizophrenia, schizoaffective disorder, bipolar disorder.
35. Tuberculosis, hepatitis B and C, HIV infection, syphilis, history or by screening.
36. Conditions after surgical procedures, if less than 6 months have passed since the intervention.
37. Therapy for cognitive impairment, balance disorders, and dizziness 21 days or less prior to Visit 1-1 date.
38. Use of an irreversible MAO inhibitor within 14 days or a reversible MAO inhibitor within 1 day prior to Visit 1-1.
39. Therapy with the following drugs and drug groups: 7 days or less before screening: Selective serotonin reuptake inhibitors (SSRIs) and selective serotonin and norepinephrine reuptake inhibitors (SSRIs); Cinnarizine and/or dimenhydrinate preparations; Cytochrome P450 3A4 (Cytochrome P450 3A4, CYP3A4) inhibitors and inducers: Erythromycin, itraconazole, nefazodone, diltiazem, verapamil, etc.; Cimetidine, warfarin, phenytoin, propranolol. Monoamine oxidase inhibitors (MAOIs): concomitant use of MAO inhibitors is prohibited, as well as taking the drug earlier than 14 days after withdrawal of an irreversible MAO inhibitor, or less than 1 day after withdrawal of a reversible MAO inhibitor.
40. Presence of a history of malignant neoplasm, except in patients who have had no disease in the past 5 years, patients with completely cured basal cell skin cancer, or completely cured carcinoma in situ.
41. Decompensated somatic diseases that, in the opinion of the investigator, would prevent the patient from complying with the regimen prescribed by the study protocol, or would prevent assessment of the efficacy of therapy and compliance according to the protocol, or could skew the results of the study.
42. Decompensated neuropsychiatric diseases, including multiple sclerosis, Parkinson's disease, endogenous depression, and others, which in the opinion of the investigator would prevent the patient from complying with the regimen prescribed by the study protocol, or would prevent assessment of therapy efficacy and compliance according to the protocol, or could skew the results of the study.
43. Female patients who are pregnant or breastfeeding or planning pregnancy within the next 15 months.
44. Patients requiring prohibited concomitant medications.
45. Participation in another clinical trial within the last 3 months prior to the date of the Screening Visit.
46. Patient's unwillingness or inability to comply with protocol procedures (in the opinion of the investigator).
47. Other conditions that, in the judgment of the investigator, preclude the patient's inclusion in the study.
48. The patient is diagnosed with COVID-19 disease at the time of screening or Randomization Visit; or the presence of symptoms of acute respiratory infections or COVID-19 within 14 days prior to screening and a positive rapid test for COVID-19 at screening.

Exclusion criteria:

1. The patient's decision to discontinue participation in the study.
2. A decision by the investigator that continued participation in the study is contrary to the patient's best interests.
3. The patient is included in the study in violation of the inclusion and non-inclusion criteria.
4. A decision by the investigator's physician to exclude the patient from the study due to lack of adequate cooperation of the patient with the investigator's physician during the study.
5. Diagnosis of acute (vestibular neuronitis, acute labyrinthitis, traumatic vestibulopathy, stroke with lesions of central and peripheral vestibular structures and others) and/or episodic vestibular syndromes (benign positional paroxysmal vertigo, Meniere's disease, vestibular migraine and others), bilateral vestibulopathy.
6. Skipping taking the study drug (3 consecutive tablets or more than 6 tablets for each period of therapy).
7. Omission of the active comparator (9 consecutive tablets or more than 17 tablets per therapy period).
8. An adverse event requiring withdrawal of investigational therapy or limiting protocol procedures.
9. The need to prescribe to the patient drugs from the "Prohibited Concomitant Therapies" section.
10. Loss of communication with the patient.
11. Pregnancy.
12. Ineffectiveness of therapy (increase from baseline or no decrease in DHI total score and MVS mean score by 25% or more from baseline after another course of therapy).
13. The patient was diagnosed with COVID-19 disease during the periods of primary and repeated therapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-01-24 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Mean vertigo score (MVS) at Visit 1-3 of the Initial Treatment Phase relative to baseline at Visit 1-1 | Day 1 - Day 28±1
  Difference in MVS assessed on Visit 1-3 and 1-1 (12-item scale with score from 0 to 4 for each item; higher scores mean a worse outcome)

SECONDARY OUTCOMES:
Change in mean MVS score at Visit 1-2 of the Initial Treatment Phase relative to baseline at Visit 1-1. | Day 1 - Day 28±1
  Assessment performed using MVS (12-item scale with score from 0 to 4 for each item; higher scores mean a worse outcome)
Change in mean MVS score at Visits 2-2, 2-3, and 2-4 of the Retreatment Period compared with Visit 2-1. | Day 1 - Day 42 ±1 (retreatment period)
  Assessment performed using MVS (12-item scale with score from 0 to 4 for each item; higher scores mean a worse outcome)
Change in mean MVS score at the visit of completion of study participation compared with the score at Visit 1-1 in patients who completed the study according to the protocol (PP(response)). | Day 1 - Day 28±1
  Assessment performed using MVS (12-item scale with score from 0 to 4 for each item; higher scores mean a worse outcome)
Percentage of patients with a ≥50% reduction in total DHI score on Visit 1-3 of the Initial Treatment Phase relative to Visit 1-1. | Day 1 - Day 28±1
  Assessment performed using DHI (25-item self-report questionnaire with total score from 0 to 100; higher scores mean a worse outcome)
Percentage of patients with a ≥50% reduction in total DHI score on Visits 2-3 and 2-4 of the Retreatment Period relative to Visit 2-1. | Day 1 - Day 42 ±1 (retreatment period)
  Assessment performed using DHI (25-item self-report questionnaire with total score from 0 to 100; higher scores mean a worse outcome)
Percentage of patients with a ≥25% reduction in total DHI score on Visit 1-3 of the Initial Treatment Phase relative to Visit 1-1. | Day 1 - Day 28±1
  Assessment performed using DHI (25-item self-report questionnaire with total score from 0 to 100; higher scores mean a worse outcome)
Percentage of patients with a ≥25% reduction in total DHI score on Visits 2-3 and 2-4 of the Retreatment Period relative to Visit 2-1. | Day 1 - Day 42 ±1 (retreatment period)
  Assessment performed using DHI (25-item self-report questionnaire with total score from 0 to 100; higher scores mean a worse outcome)
Change in total score on the DHI at Visit 1-3 of the Initial Treatment Phase compared with Visit 1-1. | Day 1 - Day 28±1
  Assessment performed using DHI (25-item self-report questionnaire with total score from 0 to 100; higher scores mean a worse outcome)
Change in total score on the DHI at Visits 2-3 and 2-4 of the Retreatment Period compared with Visit 2-1. | Day 1 - Day 42 ±1 (retreatment period)
  Assessment performed using DHI (25-item self-report questionnaire with total score from 0 to 100; higher scores mean a worse outcome)
Change in total score on the DHI at the end-of-study visit compared to the score at Visit 1-1 in patients who completed the study according to the protocol (PP(response)). | Day 1 - Day 28±1
  Assessment performed using DHI (25-item self-report questionnaire with total score from 0 to 100; higher scores mean a worse outcome)
Change in digital rating scalescore from Visit 1-1 to Visits 1-2 and 1-3 in the Primary Treatment Period. | Day 1 - Day 28±1
  Assessment performed using digital rating scale (from minimum of 0 to maximum of 10 points; higher scores mean a worse outcome)
Change in digital rating scale score from Visit 2-1 to Visits 2-2, 2-3, and 2-4 in the Retreatment Period. | Day 1 - Day 42 ±1 (retreatment period)
  Assessment performed using digital rating scale (from minimum of 0 to maximum of 10 points; higher scores mean a worse outcome)
Assessment of quality of life in patients with autonomic dysfunction syndrome accompanied by functional vertigo using the EQ-5D questionnaire at Visit 1-3 of the Initial Treatment Phase. | Day 1 - Day 28±1
  Assessment performed using EQ-5D questionnaire (5-item self-report questionnaire with total score from 0 to 100; higher scores mean a better outcome)
Assessment of quality of life in patients with autonomic dysfunction syndrome accompanied by functional vertigo using the EQ-5D questionnaire at Visits 2-3 and 2-4 of the Retreatment Period. | Day 1 - Day 42 ±1 (retreatment period)
  Assessment performed using EQ-5D questionnaire (5-item self-report questionnaire with total score from 0 to 100; higher scores mean a better outcome)
Change in total score on the Hamilton Anxiety Rating Scale HARS at Visit 1-3 of the Primary Treatment Period compared with Visit 1-1. | Day 1 - Day 28±1
  Assessment performed using HARS (21-item scale with total score from 0 to 56; higher scores mean a worse outcome)
Change in total score on the Hamilton Anxiety Rating Scale HARS at Visits 2-3 and 2-4 of the Retreatment Period compared with Visit 2-1. | Day 1 - Day 42 ±1 (retreatment period)
  Assessment performed using HARS (21-item scale with total score from 0 to 56; higher scores mean a worse outcome)
Change in VSS-SF total score at Visit 1-3 of the Initial Treatment Phase relative to baseline at Visit 1-1. | Day 1 - Day 28±1
  Assessment performed using VSS-SF score (15-item scale with score from 0 to 4 for each item; higher scores mean a worse outcome)
Change in VSS-SF total score at Visits 2- 3 and 2-4 of the Retreatment Period compared with Visit 2-1. | Day 1 - Day 42 ±1 (retreatment period)
  Assessment performed using VSS-SF score (15-item scale with score from 0 to 4 for each item; higher scores mean a worse outcome)
Change in VSS-SF total score at the end-of-study visit compared with the score at Visit 1-1 in patients who completed the study according to protocol (PP(response)). | From Day 1 to the end of the study
  Assessment performed using VSS-SF score (15-item scale with score from 0 to 4 for each item; higher scores mean a worse outcome)
Evaluation of therapy efficacy on the CGI-i scale by the patient at Visits 1-2 and 1-3 in the Initial Treatment Phase. | Day 1 - Day 28±1
  Assessment performed using CGI-i scale (scale from 0 to 7; higher scores mean a worse outcome)
Evaluation of therapy efficacy on the CGI-i scale by the physician at Visits 1-2 and 1-3 in the Primary Therapy Period. | Day 1 - Day 28±1
  Assessment performed using CGI-i scale (scale from 0 to 7; higher scores mean a worse outcome)
Evaluation of therapy efficacy on the CGI-i scale by the patient at Visits 2-2, 2-3, and 2-4 in the Retreatment Period. | Day 1 - Day 42 ±1 (retreatment period)
  Assessment performed using CGI-i scale (scale from 0 to 7; higher scores mean a worse outcome)
Evaluation of the effectiveness of therapy on the CGI-i scale by the physician at Visits 2-2, 2-3, 2-4 in the Re-Treatment Period. | Day 1 - Day 42 ±1 (retreatment period)
  Assessment performed using CGI-i scale (scale from 0 to 7; higher scores mean a worse outcome)
Proportion of patients with exacerbation (relapse) of the disease after treatment in the Primary Treatment Period during the entire follow-up period (until the visit of completion of participation in the study) | From Day 1 to the end of the study
  An exacerbation (relapse) is defined as a total DHI score ≥ 31 points
Duration of remission period after treatment in the Initial Treatment Phase. Remission means absence of episodes of exacerbations (relapses) | From Day 1 to the end of the study
  The duration of the remission period is the time from the day of completion of primary therapy to the day of the visit confirming an exacerbation (relapse) or to the day of completion of the study (if there is no exacerbation (relapse))
Clinically significant abnormalities on physical and/or neurologic examination | Day 1 - Day 28±1 (primary treatment period), Day 1 - Day 42 ±1 (retreatment period)
  Number and percentage of patients with clinically significant abnormalities found during physical and/or neurologic examination
Adverse events (AEs) | Day 1 - Day 28±1 (primary treatment period), Day 1 - Day 42 ±1 (retreatment period)
  Frequency of AEs for all treatment periods stratified by severity and frequency
Serious adverse events (SAEs) | Day 1 - Day 28±1 (primary treatment period), Day 1 - Day 42 ±1 (retreatment period)
  Frequency of SAEs
Adverse reactions | Day 1 - Day 28±1 (primary treatment period), Day 1 - Day 42 ±1 (retreatment period)
  Frequency of AEs and SAEs associated with the use of investigational drugs
Рatients with at least one AE | Day 1 - Day 28±1 (primary treatment period), Day 1 - Day 42 ±1 (retreatment period)
  Proportion of patients with at least one AE registered
Patients discontinued due to AE | Day 1 - Day 28±1 (primary treatment period), Day 1 - Day 42 ±1 (retreatment period)
  Percentage of patients who discontinued treatment due to the occurrence of AE

CONTACTS AND LOCATIONS:
Locations (4):
- Russia (4):
  - Central Clinic LLC, Bryansk
  - Federal State Budgetary Educational Institution of Higher Education "Kirov State Medical University" of the Ministry of Healthcare of the Russian Federation, Kirov
  - State Budgetary Institution of Healthcare of the City of Moscow "V.P. Demikhov City Clinical Hospital of the Department of Healthcare of the City of Moscow", Moscow
  - Private Healthcare Institution "Clinical Hospital "RZD-Medicine" of the city of Smolensk", Smolensk

IPD SHARING:
Plan to Share IPD: Undecided